CLINICAL TRIAL: NCT01427491
Title: A Prospective, Multi-center, Randomized, Comparative Clinical Study to Compare Aquacel® Ag vs. Mepilex® Border Ag to Manage Bioburden in Leg Ulcers.
Brief Title: Compare Aquacel® Ag Versus Mepilex® Border Ag to Manage Bioburden in Leg Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CW-0142-11-U358
Record Dates: First submitted 2011-08-23; First posted 2011-09-01 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Leg Ulcers
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aquacel® Ag (Active Comparator)
  Interventions: Device: Aquacel® Ag
- Mepilex® Border Ag (Active Comparator)
  Interventions: Device: Mepilex® Border Ag

INTERVENTIONS:
Device: Aquacel® Ag — Dressing will be changed during the clinic visit on day 3, 7 and 14. In between the clinic visits the dressing should be changed when needed depending on the clinical condition of the wound and the volume of exudate.
  Arms: Aquacel® Ag
Device: Mepilex® Border Ag — Dressing will be changed during the clinic visit on day 3, 7 and 14. In between the clinic visits the dressing should be changed when needed depending on the clinical condition of the wound and the volume of exudate.
  Arms: Mepilex® Border Ag

SUMMARY:
The purpose of this study is to compare the ability of Aquacel® Ag and Mepilex® Border Ag to manage bioburden in leg ulcers over a two week study period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Willing and able to provide written informed consent
* Leg ulcer will be of size ranging between 10 cm2 - 40 cm2 with moderate or heavy exudate
* Leg ulcer will exhibit at least 2 of the 4 following clinical signs: pain between 2 dressing changes, peri-ulcer skin erythema, oedema, foul odour

Exclusion Criteria:

* Known skin sensitivity to any component of the products being tested
* Subjects who have had current local or systemic antibiotics and/or topical antimicrobials applied in the week prior to inclusion
* Depth of ulcer classified as superficial (not involving dermis) or deep (exposing muscle and tendon)
* Any other medical condition which, according to the investigator, justifies the subject's exclusion from the study
* Participated in a clinical study within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Microbial load reduction | Days 1 and 14
  The relative reduction from baseline in microbial load (bio-burden) over a 2 week study period as measured by quantitative and qualitative microbiology methods.

SECONDARY OUTCOMES:
clinical evolution of the wound (presence of each of the selected clinical signs) | Days 1, 3, 7, 14
  Study's clinical signs: level of exudate (moderate or heavy at baseline), pain between 2 dressing changes, peri-ulcer skin erythema, oedema, foul odour
Occurrence of adverse events | Day 1-14

CONTACTS AND LOCATIONS:
Overall Officials: Keith Harding, Principal Investigator — Cardiff University
Locations (3):
- United Kingdom (3):
  - The Willows Centre for Health Care, Weaste, Salford
  - Wound Healing Research Unit, Cardiff University, Cardiff, Wales
  - Arrowe Park Hospital, Upton, Wirral